CLINICAL TRIAL: NCT05372978
Title: Cash Transfers for People Experiencing Homelessness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Foundations for Social Change (Unknown)
Responsible Party: Principal Investigator, Jiaying Zhao, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-02584
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Homelessness; Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to condition (cash vs control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cash (Experimental): Participants will receive a one-time unconditional cash transfer of $8,500 CAD.
  Interventions: Behavioral: Cash transfer
- Control (No Intervention): Participants will not receive a cash transfer.

INTERVENTIONS:
Behavioral: Cash transfer — Participants will receive a one-time unconditional cash transfer of $8,500.
  Arms: Cash

SUMMARY:
The primary goal of the study is to determine the impacts of a one-time unconditional cash transfer on the well-being of people experiencing homelessness.

DETAILED DESCRIPTION:
The goal of this project is to examine the effect of cash-transfers for people experiencing homelessness in Metro Vancouver. In partnership with Foundations for Social Change, we will distribute a one-time unconditional cash transfer of $8,500 to each of the 200 participants, with 200 additional participants in a control group who will not receive the cash transfer. To evaluate the effect of the cash transfer, participants will complete surveys 1, 2, 3, 6, 9, and 12 months after the cash transfer, and we will track important life outcomes such as housing, employment, health, cognitive function, and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be homeless at the time of recruitment.
2. Participants must be between 18 and 65 years of age, inclusive.
3. Participants must be a Canadian citizen or permanent resident in Canada

Exclusion Criteria:

The following participants will be excluded:

1. Participants who report severe problematic substance use (score ≥ 6 on DAST).
2. Participants who report severe problematic alcohol use (score ≥ 20 on AUDIT).
3. Participants who report severe psychiatric symptoms (score above 2 on item 5 or above 4 on items 13 or 14 on CSI).
4. Participants who report problematic gambling behavior (score ≥ 8 on PGSI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Stable housing | 1-3 months
  Number of days spent in stable housing.
Homelessness | 1-3 months
  Number of days spent homeless.
Savings | 1-3 months
  Total value of financial assets.
Total Spending | 1-3 months
  Amount of money spent on regular and one-time purchases.
Spending on Rent | 1-3 months
  Amount of money spent on rent.
Spending on temptation goods | 1-3 months
  Amount of money spent on temptation goods, such as drugs, alcohol, and cigarettes.
Cost of shelter use | 1-3 months
  Estimated societal cost of shelter use based on number of days staying in shelter

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share non-identifiable data privately with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after data collection has ended and after the data have been cleaned.